CLINICAL TRIAL: NCT01546896
Title: Effects of Buspar on Depressive Symptom Improvement and Neuroprotection in Patients With Anxiety Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, MD, PhD, MMS, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bsp2010
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- buspirone+alprazolam (Experimental)
  Interventions: Drug: buspirone+alprazolam
- alprazolam (Active Comparator)
  Interventions: Drug: alprazolam
- healthy controls (No Intervention)

INTERVENTIONS:
Drug: buspirone+alprazolam — day 1~7: buspirone 10mg/d + alprazolam 0.5mg / day 8~28: buspirone 20mg/d + alprazolam 0.5mg / day 29~56: buspirone 20~30mg/d + alprazolam 0.5mg
  Arms: buspirone+alprazolam
Drug: alprazolam — 0.5mg/d
  Arms: alprazolam

SUMMARY:
This research aims to investigate the efficacy and safety of buspirone in treating generalized anxiety disorder with depressive symptoms and to evaluate its neuroprotective effects using magnetic resonance imaging.

ELIGIBILITY:
Patient Inclusion Criteria:

* Men and women aged between 20 and 65
* Diagnosis of generalized anxiety disorder as assessed by Structured Clinical Interview for DSM-IV (SCID-IV)
* Depressive symptom scores measured by Hamilton Depression Rating Scale at screening and baseline assessments: >=8 and <=16

Healthy Control Subject Inclusion Criteria

* Healthy men and women aged between 20 and 65

Exclusion Criteria:

* Presence of any major physical or neurological illness (e.g.， head trauma, epilepsy， seizure， stroke， cerebral tumor， multiple sclerosis，cerebrovascular disease， narrow-angle glaucoma， drug hypersensitivity， etc.)
* Drug abuse in past 3 months
* Contraindications to magnetic resonance imaging (e.g., pacemaker implantation，claustrophobia, etc.)
* Diagnosis of any Axis I disorder other than generalized anxiety disorder or presence of symptoms requiring hospitalization
* Major depressive episode during past 12 months
* Depressive symptom scores measured by Hamilton Depression Rating Scale: >=17
* Women who are pregnant, breastfeeding, or planning pregnancy
* Contraindications to drugs used in the study (e.g., allergy, intolerance, etc.)
* Unstable medical illness or severe abnormality in laboratory test at screening assessment
* Use of psychoactive medications that may affect brain imaging findings
* Intelligence quotient below 80

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
change from baseline in depressive symptom scores at 8 weeks | baseline and at 8 weeks
change from baseline in depressive symptom scores at 4 weeks | baseline and at 4 weeks
change from baseline in depressive symptom scores at 1 week | baseline and at 1 week
change from baseline in anxiety symptom scores at 8 weeks | baseline and at 8 weeks
change from baseline in anxiety symptom scores at 4 weeks | baseline and at 4 weeks
change from baseline in anxiety symptom scores at 1 week | baseline and at 1 week

SECONDARY OUTCOMES:
changes from baseline in brain structure, function, and biochemical metabolism, analyzed using the computational approach | baseline and at 8 weeks
number of participants with adverse events | 8 weeks
number of participants with adverse events | 4 weeks
number of participants with adverse events | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea